CLINICAL TRIAL: NCT01933061
Title: A Randomized, Open Label, Multi-center Phase 2 Study of Nab-Paclitaxel Versus Epigenetic Modifying Therapy of CC-4386 With Nab-Paclitaxel in Subjects With Chemotherapy naïve Metastatic Melanoma
Brief Title: Study to Determine Efficacy and Safety of CC-486 With Nab-Paclitaxel Versus Nab-Paclitaxel in Patients With Chemotherapy naïve Metastatic Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic decision not to proceed with the opening of this study. There are no concerns over the safety or quality of the investigational products involved.
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-486-MEL-001
Record Dates: First submitted 2013-08-28; First posted 2013-08-30 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Metastatic Melanoma
Keywords: Skin cancer, Melanoma
MeSH Terms: conditions — Melanoma | interventions — Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abraxane 150 mg/m² Intravenous (IV) (Experimental)
  Interventions: Drug: Abraxane
- CC-486 orally plus Abraxane IV (Experimental)
  Interventions: Drug: Abraxane

INTERVENTIONS:
Drug: Abraxane — Abraxane 150- mg/m² IV on Days 1, 8, and 15 of a 28-day cycle
  Other Names: nab-paclitaxel, ABI-007
  Arms: Abraxane 150 mg/m² Intravenous (IV)
Drug: Abraxane — Abraxane 150 mg/m^2 intravenously on Days 1, 8, and 15 of a 28-day cycle
  Other Names: nab-paclitaxel, ABI-007
  Arms: CC-486 orally plus Abraxane IV

SUMMARY:
A phase 2, open-label randomized, multicenter trial to compare CC-486 in combination with Abraxane administered weekly with respect to overall survival, objective tumor response rate and Progression-Free Survival (PFS) in participants diagnosed with metastatic malignant melanoma.

DETAILED DESCRIPTION:
The study will consist of the following phases:

* Screening (Baseline) Assessments: Performed within 21 days of randomization.
* Randomization: Subjects will be randomized within 21 days of starting their Baseline assessments.
* Treatment: Therapy may continue in the absence of clinically significant disease progression and unacceptable toxicity.
* Response Assessments: Subjects will be evaluated by investigators for CR, PR, stable or progressive disease every 6 weeks from the start of treatment until progressive disease is documented.

Responders and subjects with stable disease (SD) should continue on study unless they develop unacceptable toxicity, they start a new anticancer therapy, withdrawal of consent, physician decision or death.

* End of Study (EOS)/Treatment Evaluation: At the time subjects are removed from study, laboratory and clinical evaluations will be performed.
* Follow-up for Disease Progression:

  - Subjects who stop treatment prior to developing disease progression should be followed without further treatment until progressive disease is documented or until the treating physician feels additional treatment is required.
* Follow-up for Survival:

  * Post study, subject survival status will be monitored on a monthly basis for 6 months from discontinuation from the study and every 3 months thereafter, until death or study termination in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically or cytologically confirmed cutaneous BRAF wild-type malignant melanoma with evidence of metastasis (Stage IV).

  2. No prior cytotoxic chemotherapy for metastatic malignant melanoma is permitted. No prior adjuvant cytotoxic chemotherapy is permitted.
  * Up to one prior regimen with the following classes of agents is permitted:

    o Targeted biologic agents (e.g. interleukin 2 [IL-2], granulocyte macrophage colony stimulating factor [GM-CSF], other cytokines or unarmed monoclonal antibodies)

    o Targeted small molecule inhibitors (e.g., kinase inhibitors, heat shock protein [HSP] inhibitors, etc.).
    * Immune checkpoint inhibitors (e.g. anti-CTLA4, anti-PD1, anti-PD-L1).
    * Prior adjuvant therapy with interferon and/or vaccines is permitted.
  * Prior treatments should be completed 4 weeks prior to enrollment in the study (ie, randomization).

    3. Male or non-pregnant and non-lactating female, and ≥ 18 years of age at the time of signing the informed consent document.
  * If heterosexually active, the subject must agree to use medical doctor-approved contraception throughout the study, and for 6 months after last dose of study drug.

    4. History of malignancy in the last 5 years; subjects with prior history of in situ cancer or basal or squamous cell skin cancer are eligible.
  * Subjects with other malignancies are eligible if they were cured by surgery (with or without radiotherapy) and have been continuously disease-free for at least 5 years.

    5. Radiographically-documented measurable disease (defined by the presence of at least one radiographically documented measurable lesion including measurable cutaneous metastasis).

    6. Adequate haemtological and biochemical parameters:
  * ANC ≥ 1.5 x 109 cells/L.
  * Platelets ≥ 100 x 109 cells/L.
  * Hgb ≥ 9 g/dL.
  * AST (SGOT) or ALT (SGPT) ≥ 2.5x upper limit of normal range (ULN);

    o ≤ 5.0 x ULN if hepatic metastases present.
  * Total bilirubin ≤ ULN. Creatinine ≤ 1.5 mg/dL. 8. ECOG performance status 0 to 1.

Exclusion Criteria:

* 1. History of or current evidence of symptomatic brain metastases (brain Computed Tomography (CT)/Magnetic Resonance Imaging (MRI) is needed to exclude brain metastasis), including leptomeningeal involvement.

  2. Subject has pre-existing peripheral neuropathy of National Cancer Institute NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) Scale of Grade ≥ 2.

  3. Prior radiation to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 months
  PFS is defined as the time from randomization date to disease progression according to RECIST response guideline

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 24 months
  OS is defined as the time from the date of randomization to the date of death.
PFS | Up to 24 months
  PFS based on investigator assessment; PFS is defined as the time from randomization date to disease progression according to RECIST response guideline
Objective Response Rate (ORR) | Up to 24 months
  Number (%) of subject who achieve an objective complete or partial response.
Disease Control Rate (DCR) | Up to 24 months
  Number (%) of subject with Stable Disease (SD) ≥ for 18 weeks or complete or partial response.
Safety | Up to 24 months
  Incidence and severity of Adverse events (AE) will be analyzed in terms of treatment-emergent AEs defined to be any AE that begin or worsen in severity after study drug initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Hege, MD, Study Director — Celgene Corporation